CLINICAL TRIAL: NCT04254666
Title: A Pilot and Feasibility Study to Promote Physical and Food Literacy Among Children With Intellectual Disabilities
Brief Title: New Skills - No Scores Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Massachusetts, Boston (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Carol Curtin, PhD, Professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H00017816; 1R21HD099435-01 (NIH)
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Intellectual Disability
Keywords: physical literacy; food literacy
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Literacy & Food Literacy Intervention (Other): This is a pilot project to assess the feasibility of a physical literacy and food literacy intervention for adolescents with ID ages 12-16 years.
  Interventions: Behavioral: Physical Literacy & Food Literacy Intervention.

INTERVENTIONS:
Behavioral: Physical Literacy & Food Literacy Intervention. — A 12-week intervention designed to expose adolescents with ID to a variety of sports skills and healthy eating concepts to equip them with skills and confidence to participate in sports and make healthy food choices. The program will follow a protocol adapted to meet the needs of a diverse group of children with ID. Sessions will be held 1 time/week for 75 minutes virtually; 35 minutes will focus on sport skills activities with 35 minutes devoted to healthy eating.
  Other Names: New Skills - No Scores

SUMMARY:
The purpose of this study is to test the feasibility of a physical literacy and food literacy intervention for children with Intellectual Disabilities ages 12-16 years. The Investigators plan to assess preliminary efficacy of the intervention for increasing 1) physical literacy including movement skills, physical self-concept, and desire to participate in physical activity and 2) food literacy including knowledge around making healthy food choices, basic food preparation skills, and engaging in healthy eating behavior.

DETAILED DESCRIPTION:
Children with intellectual disabilities (ID) are more likely than typically developing children to have higher cardio-metabolic risk factors, lower levels of health-related fitness, and be overweight and obese. As such, they represent a health disparities population. Low physical activity levels, increased sedentary time, and poor diet quality are likely contributors to these inequities. The goal of the Investigators is to develop strategies that enable children with ID to attain optimal health by meeting US Physical Activity Guidelines and Dietary Guidelines for Americans. To achieve this goal, children with ID must develop physical literacy and food literacy - the knowledge, skills, confidence and desire to participate in physical activity and make healthy food choices. This project seeks to:1) test the feasibility of a physical literacy and food literacy intervention for children with ID, and 2) preliminarily assess the efficacy of the intervention for increasing physical literacy including movement skills, confidence, and desire to participate in physical activity, and food literacy including knowledge around making healthy food choices, basic food preparation skills, and engaging in healthy eating behavior. Thirty male (n=15) and female (n=15) children with ID ages 12-16 will participate in a 12-week , virtual, combined sport skills sampling and healthy eating education program. Weekly online sessions will include 35 minutes of sports skills activities and 35 minutes of educational and skill activities to promote healthy eating. Sport skill sampling activities will aim to develop locomotor and object control skills via four 3-week sessions including dribbling, locomotor skills, ball skills, and a fourth session combining them all. Healthy eating sessions will focus on increasing knowledge to identify healthy foods and to make healthy choices, basic skills for preparing food, and a taste test thematically related to the lesson. The intervention will also include a practice component called "Give it Try." Children will be provided with a piece(s) of sports equipment (e.g., soccer ball, basketball) and skill videos with instructions and fun ideas for practicing sport skills outside of program sessions, additionally as part of "Give it a Try" we encourage participants to try new foods outside of the intervention. Process measures of demand, acceptability, and implementation will be obtained to test feasibility, and a pre-test/post-test design will allow for preliminary data on efficacy of the intervention. Measures of physical literacy include the Test of Gross Motor Development, 3rd ed, Physical Self-Inventory-ID, and Children's Self- Perceptions of Adequacy in and Predilection for Physical Activity scale. Measures of food literacy include a questionnaire on food knowledge and parent proxy report of dietary patterns based on a modified food frequency questionnaire (FFQ), and questions from the Youth Risk Behavioral Surveillance Survey. This early phase study is a step toward promoting health and reducing the inequities that exist for children with ID.

ELIGIBILITY:
Inclusion Criteria:

* measured IQ and adaptive functioning scores of ≤75 as measured by the Kaufman Brief Intelligence Test-2 (KBIT-2) and Vineland Adaptive Behavior Scales-III (VABS-III). A score > 75 for participants that do not have a syndrome that is associated with ID will be exclusionary. However, participants with such syndromes (e.g., Down syndrome) may have scores above this cut-point but are still classified as having an intellectual disability and thus will qualify for the study.
* Participants must be ambulatory and in sufficiently good health to engage in moderate-to-vigorous physical activity
* able to communicate verbally in English, follow simple instructions, and provide assent.
* approval from the participants' primary care physician and specialists (as necessary) will be required for participation.

Exclusion Criteria:

* uncontrolled medical or significant psychiatric condition
* insulin-dependent diabetes
* physical/orthopedic impairment that would preclude participation in physical activity
* legally blind or deaf
* habitual problem behaviors such as aggression, noncompliance, or leaving an activity area.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Curtin, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share data from this pilot project.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Literacy & Food Literacy Intervention
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: adolescents with intellectual disabilities
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Motivation and Confidence in Physical Activity
Description: Physical Self-Concept will be measured using the Very Short Form of the Physical Self-Inventory-Intellectual Disability (PSI-VSF-ID). The PSI-VSF-ID is a 12-item questionnaire that measures six dimensions of self-concept: 1) Global Self-Concept; 2) Physical Self-Worth; 3) Sport Competence; 4) Physical Attractiveness; 5) Physical Condition; and 6) Physical Strength. Four response options range from "very true" to "not at all true", and a visual answer scale uses smiling/frowning faces effective for use with adolescents with ID. Higher scores indicate higher self-concept in the aforementioned domains. We will examine changes in participants' physical self-concept between baseline and post-intervention.
Time Frame: Baseline and Post intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
score on a scale
  Baseline - Global Self-concept (Range: 0 - 4) | 3.42 (0.74)
  Post Intervention - Global Self-concept (Range: 0 - 4) | 3.42 (0.80)
  Baseline - Physical Self-worth (Range: 0 - 4) | 3.17 (0.98)
  Post Intervention - Physical Self-worth (Range: 0 - 4) | 3.42 (0.92)
  Baseline - Physical Condition (Range: 0 - 4) | 2.50 (1.26)
  Post Intervention - Physical Condition (Range: 0 - 4) | 2.75 (0.69)
  Baseline - Sport Competence (Range: 0 - 4) | 2.92 (0.80)
  Post Intervention - Sport Competence (Range: 0 - 4) | 3.33 (0.52)
  Baseline - Physical Attractiveness (Range: 0 - 4) | 3.08 (0.66)
  Post Intervention - Physical Attractiveness (Range: 0 - 4) | 3.17 (0.88)
  Baseline - Physical Strength (Range: 0 - 4) | 2.92 (0.86)
  Post Intervention - Physical Strength (Range: 0 - 4) | 3.17 (0.68)

2. Primary Outcome: Movement/Motor Skills
Description: Movement/Motor Skills will be assessed using the Test of Gross Motor Development (3rd ed). The TGMD-3 assesses 13 fundamental motor skills related to 1) locomotor skills and 2) ball skills. The TGMD-3 is a direct observation skill assessment with 3-5 performance criteria for each skill. We will assess: skipping, two-foot jumping, one-foot hopping, sideways sliding, overhand throw, underhand throw, catch, hand dribble, and kick. The TGMD-3 will be administered via Zoom at baseline and post-12 weeks.A trained professional will review and code the video-recorded TGMD-3 performance on each skill and provide a score at baseline and post-test. For all of the ranges higher scores equal greater motor proficiency.
Time Frame: Baseline and Post intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
score on a scale
  Baseline - Total Motor Skills (Range: 0 - 66) (higher indicate better motor skills) | 24.0 (10.6)
  Post Intervention - Total Motor Skills (Range: 0 - 66) | 27.8 (14.2)
  Baseline - Locomotive Skills (Range: 0 - 30) | 7.8 (6.4)
  Post Intervention - Locomotive Skills (Range: 0-30) | 7.7 (5.5)
  Baseline - Hop (Range: 0 - 8) | 2.17 (1.83)
  Post Intervention - Hop (Range: 0 - 8) | 2.5 (2.17)
  Baseline - Skip (Range: 0 - 6) | 1.33 (2.07)
  Post Intervention - Skip (Range: 0 - 6) | 0.66 (1.03)
  Baseline - Jump (Range: 0 - 8) | 2.67 (1.51)
  Post Intervention - Jump (Range: 0 - 8) | 2.83 (2.48)
  Baseline - Slide (Range: 0 - 8) | 1.67 (1.03)
  Post Intervention - Slide (Range: 0 - 8) | 1.67 (0.82)
  Baseline - Ball Skills (Range: 0 - 36) | 16.2 (7.1)
  Post Intervention - Ball Skills (Range: 0 - 36) | 20.2 (9)
  Baseline - Dribble (Range: 0 - 6) | 2.17 (2.14)
  Post Intervention - Dribble (Range: 0 - 6) | 3.0 (1.9)
  Baseline - Catch (Range: 0 - 6) | 5.0 (1.1)
  Post Intervention - Catch (Range: 0 - 6) | 5.0 (1.55)
  Baseline - Kick (Range: 0 - 8) | 2.0 (1.41)
  Post Intervention - Kick (Range: 0 - 8) | 2.83 (2.93)
  Baseline - Overhand Throw (Range: 0 - 8) | 1.0 (1.67)
  Post Intervention - Overhand Throw (Range: 0 - 8) | 1.83 (2.48)
  Baseline - Underhand Throw (Range: 0 - 8) | 3.67 (3.14)
  Post Intervention - Underhand Throw (Range: 0 - 6) | 4.83 (1.94)

3. Primary Outcome: Desire to Participate in Physical Activity
Description: The adequacy and predilection for physical activity subscale of the Canadian Assessment of Physical Literacy - 2nd Ed (CAPL-2) Questionnaire estimates the participant's desire to participate in physical activity. The 6-item questionnaire subscale includes 3 items that assess perceived adequacy (i.e., self-perception that one has the capability to achieve an acceptable standard of success conceptualized by the self and others) and 3 items that assess perceived predilection for physical activity (i.e., likelihood of selecting physical activity over sedentary behavior when given the choice). This is a shortened and refined version of the original CAPL Questionnaire. The adequacy and predilection subscale, called "What's Most Like Me?", uses an alternative response choice format to present statements about preferences and feelings about physical activity. For all ranges higher scores indicate higher levels of perceived self concept, motivation, and competency for physical activity.
Time Frame: Baseline and Post intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
score on a scale
  Baseline - Perceived Competence for PA (Range: 0 - 3) | 1.5 (1.38)
  Post Intervention - Perceived Competence for PA (Range: 0 - 3) | 2.67 (0.52)
  Baseline - Intrinsic Motivation for PA (Range: 0 - 3) | 2.0 (0.89)
  Post Intervention - Intrinsic Motivation for PA (Range: 0 - 3) | 2.67 (0.52)
  Baseline - Perceived Adequacy for Sports and Active Games (Summed score; Range: 0 - 6) | 4.17 (1.94)
  Post Intervention - Perceived Adequacy for Sports and Active Games (Summed score; Range: 0 - 6) | 4.67 (1.86)

4. Primary Outcome: Healthy Food Knowledge.
Description: Will be measured with a hands-on Food Knowledge/Skills test adapted from knowledge tests for typically developing children and children with ID developed by the investigative team. Participants will be asked to classify individual foods into food groups (e.g., an apple belongs in the fruit group), and other healthy eating concepts such as identifying whole grains, choosing the healthiest meal between two pictures of plates with food on them, and identifying beverages that have less sugar. For each item, answers will be scored as correct or incorrect (0 or 1) or "I don't know" (0) and summed for a total of percent correct. We will examine changes in participants' food knowledge/skills between baseline and post-intervention. Higher scores indicate increased knowledge.
Time Frame: Baseline and Post intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
score on a scale
  Baseline - Identifying Whole Grain Foods (Range: 0 - 5) | 3.17 (0.75)
  Post Intervention - Identifying Whole Grain Foods (Range: 0 - 5) | 3.33 (0.82)
  Baseline - Identifying Drinks with Less Sugar (Range: 0 - 2) | 1.5 (0.84)
  Post Intervention - Identifying Drinks with Less Sugar (Range: 0 - 2) | 1.83 (0.41)
  Baseline - Identifying the Healthier Meal (Range: 0 - 2) | 1.33 (1.03)
  Post Intervention - Identifying the Healthier Meal (Range: 0 - 2) | 1.83 (0.41)
  Baseline - Identifying the Healthier Snack (Range: 0 - 3) | 2.33 (1.03)
  Post Intervention - Identifying the Healthier Snack (Range: 0 - 3) | 2.33 (1.21)

5. Primary Outcome: Foods Participant is Willing to Eat
Description: To assess teens' willingness to eat specific foods, parents completed a modified Food Frequency Questionnaire that contained a list of 108 common foods to report their teen's willingness to eat various food items ("no, my teen will not eat this" and "yes, my teen will eat this"). Parents who reported that they have not served the food item to their child were coded as missing. Parent responses were dichotomized to indicate teen willingness to eat the food and summed within their respective food groups (vegetables, fruits, proteins, grains, and dairy).
  The mean number of foods for each food group was used for analysis. Higher values indicate an increase in the participants' willingness to eat the foods in the specified food group.
Time Frame: Baseline and Post intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: number of foods in food group
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
number of foods in food group
  Baseline - Vegetables (mean) | 20.83 (4.58)
  Post Intervention - Vegetables (mean) | 23.5 (4.81)
  Baseline - Fruits (mean) | 16.17 (4.67)
  Post Intervention - Fruits (mean) | 17.00 (4.43)
  Baseline - Proteins (mean) | 13.83 (1.94)
  Post Intervention - Proteins (mean) | 14.83 (1.60)
  Baseline - Grains (mean) | 11.50 (1.64)
  Post Intervention - Grains (mean) | 13.17 (1.17)
  Baseline - Dairy (mean) | 3.50 (0.55)
  Post Intervention - Dairy (mean) | 3.83 (0.41)
Statistical Analysis 1: Comparison: Physical Literacy & Food Literacy Intervention; Test type: Other; pre and post scores for this measure are presented as the percent of foods correctly classified

6. Primary Outcome: Food Categorization
Description: Participants will be asked to classify individual foods into food groups (e.g., an apple belongs in the fruit group). For each item, answers are scored as correct or incorrect (0 or 1) or "I don't know" (0) and summed for a total of percent correct. Higher percentage scores indicate increased ability to classify foods correctly. Range is 0-100%.
Time Frame: Baseline and Post Intervention (within 1 month)
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
percent correct
  Baseline Categorization of food into food groups (% Correct) | 64.7 (47.8)
  Post Intervention Categorization of food into food groups (% Correct) | 79.3 (40.5)

7. Secondary Outcome: Participant (Teen) Enjoyment and Satisfaction
Description: Will be measured with a survey of enjoyment, satisfaction, and perceived appropriateness of key elements of the program. Survey will include closed-ended questions with Likert scale response categories, and will be verbally administered.
Time Frame: Week 12
Measure: Number; unit: % participants indicating agreement
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
% participants indicating agreement
  Percent reporting liking the sport skills part of the program | 100
  percent reporting liking the sports skills practice between sessions | 50
  percent reporting liking the nutrition education | 83
  percent reporting liking the taste tests | 83
  percent reporting liking trying two new foods each week | 100
  percent reporting that the sports skills were just right | 83
  percent reporting the nutrition education sessions were just right | 83

8. Secondary Outcome: Parent Satisfaction
Description: Will be measured with a survey of satisfaction and perceptions of the program that queries key elements of the program. Survey will include closed-ended questions with Likert scale response categories, and space for open-ended comments and feedback.
Time Frame: Week 12
Measure: Number; unit: % parents indicating agreement
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
% parents indicating agreement
  % parents reporting that program was effective in motivating their teen to eat healthy foods. | 83
  % parents reporting program was effective in increasing teens interest physical activity/sports | 50
  % parents reporting they would recommend the program to other families of teens with ID | 83
  % parents reporting overall satisfaction with the program | 83

9. Secondary Outcome: Attendance
Description: Attendance was recorded at each weekly session of the 12-week intervention. Absences and withdrawals were documented. The total % of sessions that all participants attended is reported.
Time Frame: Weekly for 12 weeks
Measure: Number; unit: % sessions the participants attended
Units Other Than Participants: total # of sessions
Arm/Group | Physical Literacy & Food Literacy Intervention
Number analyzed (Participants) | 6
Number analyzed (total # of sessions) | 72
% sessions the participants attended | 87.5

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Physical Literacy & Food Literacy Intervention
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Due to the COVID-19 Pandemic the study was halted in March of 2020 which required creating a new intervention to be delivered remotely which began in March of 2022.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT04254666/Prot_SAP_000.pdf